CLINICAL TRIAL: NCT04952922
Title: Changes to Function and Quality of Life and Patient Experience for Patients Undergoing Treatments for Recurrent Oropharyngeal Cancer
Acronym: FUNQOLR
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5242
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Oropharynx Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Therapeutics; Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment for recurrent oropharyngeal cancer (curative/ palliative) — Open salvage surgery, transoral robotic surgery, palliative chemotherapy, immunotherapy.

SUMMARY:
The purpose of this research project is to measure changes in communication, swallowing and quality of life and individual patient priorities which may happen over time in patients with a diagnosis of recurrent head and neck cancer, specifically recurrent cancer (cancer which has returned after previous treatment) of the back of the throat, the tonsils and/or the base of tongue (recurrent oropharyngeal cancer) and what it is like for patients and their significant others to experience these changes over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 years or over) competent to provide consent
* Have a diagnosis of recurrent OPC
* Have adequate linguistic and cognitive function to participate in interview
* English speaking

Exclusion Criteria:

* Any previous medical condition, other than HNC, which has a known impact on communication/ swallowing (Parkinson's Disease, Multiple Sclerosis, cerebral vascular accident (CVA)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of recurrent, residual or new primary oropharyneal cancer in a previously irradiated field.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Difficulties recruiting participants to the study, number recruited will be adequate for analysis and will meet criteria for primary endpoint
Groups:
- Group 1: Patients with a diagnosis of recurrent oropharyngeal cancer - prospective
Period: Overall Study
Arm/Group | Group 1
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 12
Age, Continuous [Median (Inter-Quartile Range); unit: YEARS] | 64 [55 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Swallowing Related Quality of Life
Description: Performance Scale for Head and Neck Cancer (PSS-HN) Normalcy of Diet (NoD) scores
  Three subscales: Normalcy of Diet, Understandability of Speech, Eating in Public
  Scores are combined to describe patient function in 6 areas (physical well-being, social and family well-being, relationship with doctor, emotional well-being, functional well-being, head & neck related symptoms)
  Total score Scale 0 -100, a higher score indicating better performance/higher quality of life
  The score reported is the combined score with the total being the sum of the sub-scale scores
Time Frame: Baseline, 3 months, 6 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1
Number analyzed (Participants) | 25
score on a scale
  Baseline | 50 [0 to 100]
  3 months | 40 [0 to 100]
  6 months | 40 [0 to 100]

2. Secondary Outcome: Swallowing Status Measured Using the 100ml Water Swallow Test
Description: The Water Swallow Test is used to monitor swallow performance and possible aspiration - patients are viewed to have failed the test if they cough, have a wet voice quality post swallow or are unable to complete the task.
Time Frame: Baseline, 3 months, 6 months
Population: Some participants were unable to complete/did not wish to complete the water swallow test
Measure: Median (Inter-Quartile Range); unit: ml/second
Arm/Group | Group 1
Number analyzed (Participants) | 17
ml/second
  Baseline | 9.7 [6.2 to 16.3]
  3 months: number analyzed (Participants) | 5
  3 months | 16.6 [13.3 to 33.2]
  6 months: number analyzed (Participants) | 5
  6 months | 17.9 [12 to 33.1]

3. Secondary Outcome: Swallowing Status Measured With the Standardisation Initiative Functional Diet Scale (IDDSI-FDS)
Description: The scale consists of 8 levels (0-7) where drinks are measured as 0-4 to describe thickness (0 being thin, 4 being extremely thick) and foods are measured as 3-7 (3 being liquidised, 7 being regular/easy to chew)
  A higher score indicates a higher level of swallowing function, 0 being the lowest score, 7 being the highest score
Time Frame: Baseline, 3 months, 6 months
Population: Not all participants completed the questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1
Number analyzed (Participants) | 25
score on a scale
  Baseline | 7 [0 to 7]
  3 months: number analyzed (Participants) | 23
  3 months | 6 [0 to 7]
  6 months: number analyzed (Participants) | 21
  6 months | 6 [0 to 7]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to 6 months
Description: All-Cause Mortality was assessed up to 6 months - no other adverse event data collected due to non-interventional nature of study
Arm/Group | Group 1
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT04952922/Prot_SAP_000.pdf